CLINICAL TRIAL: NCT03318575
Title: Safety and Effectiveness of Remote Ischemic Conditioning With the autoRIC Prior to Elective Percutaneous Coronary Intervention (PCI) Study
Brief Title: Remote Ischemic Conditioning Using the autoRIC
Acronym: SHIELD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CellAegis US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CS-000002 2013-SHIELD
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Ischemia-Reperfusion Injury
Keywords: remote ischemic conditioning (RIC); percutaneous coronary intervention; PCI; cardiac troponin I; cardiac catheterization; myocardial injury; myocardial necrosis; autoRIC; Ischemia-Reperfusion Injury (IRI); Automated Remote Ischemic Conditioning
MeSH Terms: conditions — Reperfusion Injury; Cardiomyopathy, Dilated, 1FF; Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- autoRIC (Experimental): The autoRIC device will be used on subjects randomized to the treatment group.
  Interventions: Device: autoRIC
- autoRIC Sham (Sham Comparator): The autoRIC Sham device will be used on subjects randomized to the control group.
  Interventions: Device: autoRIC Sham

INTERVENTIONS:
Device: autoRIC — Automated Remote Ischemic Conditioning
  Arms: autoRIC
Device: autoRIC Sham — Automated Remote Ischemic Conditioning Sham
  Arms: autoRIC Sham

SUMMARY:
The purpose of the study is to evaluate the hypothesis that patients receiving remote ischemic conditioning using the autoRIC device show statistically significant reduction in the prevalence of ischemia-reperfusion injury to the myocardium as compared to patients in the autoRIC Sham device arm (within 12-24 hours post non-emergent PCI with stent implantation).

DETAILED DESCRIPTION:
This is a multi-center, randomized, controlled single-blind clinical trial to evaluate the safety and effectiveness of the autoRIC device to attenuate myocardial injury as measured by cardiac Troponin I (cTnI) levels in patients undergoing PCI with stent implantation.

Eligible patients that are scheduled for an elective PCI, or unscheduled/non-emergent PCI, or patients scheduled for a diagnostic catheterization procedure with orders of "treat as indicated" will be enrolled in the study. Patients will undergo remote ischemic conditioning with the autoRIC device or the control procedure with the autoRIC Sham device completed ≤ 1 hour prior to balloon or stent inflation. Subjects will have measurements of cTnI levels at baseline and 4-8 and 12-24 hours post completion of the PCI procedure. Adverse events will be recorded through study exit for all patients. Patients will be exited from the study after completion of their 30-day post-procedure telephone follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age
2. Subject is scheduled for elective PCI, or unscheduled but non-emergent PCI, or diagnostic catheterization with PCI if indicated. For non-elective cases, there must be at least two troponin levels within the upper limit of normal (ULN), at least 6 hours apart prior to the index procedure
3. Subject is willing and capable of providing written informed consent
4. If the subject is a woman of childbearing potential, she must have had a negative pregnancy test within 24 hours of the study procedure

Exclusion Criteria:

1. Subject requires emergency PCI (i.e., PCI for evolving or ongoing STEMI/NSTEMI)
2. Subject has an elevated troponin level (cTnI or T) > ULN at baseline, based on lab results obtained from the treating institution
3. Subject is scheduled to undergo PCI with the use of Propofol
4. Subject has a recent history of drug treatment with potassium channel activators (e.g., Nicorandil) or potassium channel blockers (e.g., sulfonylureas) during the last 7 days prior to baseline
5. Subject had STEMI during the last 4 weeks prior to baseline. (Note: NSTEMI in the last 4 weeks prior to baseline is allowed if the baseline troponin is ≤ ULN.)
6. Underwent a CABG in the last 4 weeks prior to baseline
7. Had a PCI within the last 7 days prior to baseline
8. Subject has a life expectancy < 6 months
9. Subject has NYHA Class IV or decompensated heart failure
10. Subject has peripheral vascular disease requiring intervention during the index hospitalization or within 4 weeks post-procedure
11. Subject has either serum creatinine >2 times the age-appropriate upper limit of normal, a glomerular filtration rate (GFR) of < 30 mL/min/1.73m2 or requires dialysis
12. Subject has systolic blood pressure > 200 mmHg
13. Subject is currently being treated with systemic oral or I.V. steroids
14. Subject has a known bleeding disorder or known abnormality of blood flow to the limb to be treated
15. Subject has peripheral nerve injury, abnormal nerve supply, peripheral neuropathy or pre-existing traumatic injury to the limb to be treated
16. Subject is scheduled for a PCI procedure to treat a known Chronic Total Occlusion (CTO) lesion
17. Subject is currently participating in or is planning to participate in another investigational drug or device trial, prior to the 30-day follow-up visit. (Note: Observational studies or post-approval studies/ registries, are allowed.)
18. Planned (staged) post-index procedure intervention within 30 days (i.e., PCI of non-target lesions in any vessel or CABG). (Note: Planned revascularization (PCI or bypass) of a non-target lesion >30 days following the index procedure is allowed.)
19. Any cardiac surgical procedure planned within 30 days post-enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
(Primary Effectiveness) Attenuation of myocardial injury assessed by Cardiac Troponin I levels (cTnI) | 12-24 hours
  The proportion of subjects with cTnI levels above the 99th percentile Upper Reference Limit (URL) (0.04 ng/mL) 12-24 hours post-PCI.
(Primary Safety) Major Adverse Cardiac Events (MACE) | 30 days
  The proportion of subjects with major adverse cardiac events (MACE) within 30 days. MACE is defined as: death, stroke, myocardial infarction or the need for target vessel revascularization.

SECONDARY OUTCOMES:
Type 4a Myocardial Infarction (MI) | 12-24 hours
  The proportion of subjects with a Type 4a MI within 12-24 hours post- PCI.
Contrast-Induced Acute Kidney Injury (CI-AKI) | 12-24 hours
  The proportion of subjects with CI-AKI defined as > 25% or 0.5 mg/dl increase in serum creatinine above baseline within 12-24 hours post-PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Roxana Mehran, MD, Principal Investigator — Cardiovascular Medicine Associates
Locations (16):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Danbury Hospital, Danbury, Connecticut
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - Iowa Heart Center, Des Moines, Iowa
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Southside Hospital, Bay Shore, New York
  - North Shore University Hospital, Manhasset, New York
  - Mount Sinai Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Staten Island University Hospital, Staten Island, New York
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - NC Heart and Vascular Research, Raleigh, North Carolina
- Canada (2):
  - William Osler Health System, Brampton, Ontario
  - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No